CLINICAL TRIAL: NCT02558855
Title: The Effects of Thrust Joint Manipulation on the Resting and Contracting Thickness of Transversus Abdominis in Subjects With Low Back Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nova Southeastern University (Other)
Collaborators: DeRosa Physical Therapy (Unknown); University of Nevada, Las Vegas (Other)
Responsible Party: Principal Investigator, Kelly Fosberg, Principal Investigator; Nova Southeastern University PhD student in Physical Therapy, Nova Southeastern University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 01151512
Record Dates: First submitted 2015-09-22; First posted 2015-09-24 (Estimated); Last update posted 2016-04-12 (Estimated); Status verified 2016-04

CONDITIONS: Low Back Pain
Keywords: Thrust Joint Manipulation; Non-thrust Joint Manipulation; Transversus Abdominis
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Thrust Joint Manipulation (Active Comparator): Patients will receive thrust joint manipulation to their lumbar spine in side lying.
  Interventions: Other: Thrust Joint Manipulation of the Lumbar Spine
- Non-thrust Joint Manipulation (Sham Comparator): Patients will receive non-thrust joint manipulation, oscillations into slight rotation, without cavitation, to their lumbar spine in side lying.
  Interventions: Other: Non-thrust Joint Manipulation of the Lumbar Spine

INTERVENTIONS:
Other: Thrust Joint Manipulation of the Lumbar Spine
  Arms: Thrust Joint Manipulation
Other: Non-thrust Joint Manipulation of the Lumbar Spine
  Arms: Non-thrust Joint Manipulation

SUMMARY:
The primary aim of this study is to examine how different physical therapy interventions affect the resting state and contraction state of a certain abdominal muscle in patients with low back pain.

DETAILED DESCRIPTION:
Patients with low back pain (LBP) will undergo ultrasound imaging of the transversus abdominis to measure the muscle thickness at rest and at the contracted state prior to intervention and again immediately after intervention. In this randomized controlled trial, patients will be randomized into one of two groups. One group will receive the intervention of thrust joint manipulation of the lumbar spine and the other group will receive the intervention of non-thrust joint manipulation of the lumbar spine.

ELIGIBILITY:
Inclusion Criteria:

* Adults between 18-70 years of age with primary symptom of LBP, with or without referral into lower extremity.
* Subjects must be able to read and write in English.

Exclusion Criteria:

* Presence of serious pathology.
* Diagnosis of spinal stenosis or symptoms in both lower legs (changes in sensation, muscle weakness).
* Any history of low back surgery, rheumatoid arthritis, osteoporosis, osteopenia, scoliosis, or ankylosing spondylitis.
* Pregnancy
* Pending legal action.
* Prior surgery to the lumbar spine or fractures of the lumbar spine.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 67 (Actual)
Dates: Start 2015-01; Primary Completion 2015-11 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
Transversus Abdominis thickness change. | Baseline to immediately after the intervention (within 5 minutes).
  Measurement of change in thickness from resting to contraction will be compared at baseline (pre-intervention) to immediately following the intervention (post-intervention). The study is looking at the immediate effects so there is no short-term or longer follow up.

SECONDARY OUTCOMES:
Oswestry Low Back Pain Questionnaire | Baseline, immediately post-intervention (within 5 minutes), and follow-up within 48 hours over the phone.
  The score of the Oswestry Low Back Pain Questionnaire will be compared from baseline, immediately post-intervention (within 5 minutes), and follow-up within 48 hours over the phone.
Numeric Pain Rating Scale | Baseline, immediately post-intervention (within 5 minutes), and follow-up within 48 hours over the phone.
  The score of the Numeric Pain Rating Scale will be compared from baseline, immediately post-intervention (within 5 minutes), and follow-up within 48 hours over the phone.
Fear-Avoidance Beliefs Questionnaire | Baseline, immediately post-intervention (within 5 minutes), and follow-up within 48 hours over the phone.
  The score of the Fear-Avoidance Beliefs Questionnaire will be compared from baseline, immediately post-intervention (within 5 minutes), and follow-up within 48 hours over the phone.
Global Rating of Change | Immediately post-intervention (within 5 minutes) and at follow-up within 48 hours over the phone.
  The score of the Global Rating of Change will be compared from immediately post-intervention (within 5 minutes) and follow-up within 48 hours over the phone.

CONTACTS AND LOCATIONS:
Overall Officials: Kelly K Fosberg, DPT, Principal Investigator — Nova Southeastern University and DeRosa Physical Therapy; Joshua Cleland, PhD, Study Chair — Nova Southeastern University
Locations (2):
- United States (2):
  - DeRosa Physical Therapy, Flagstaff, Arizona
  - University of Nevada, Las Vegas, Las Vegas, Nevada

REFERENCES:
- [Derived] Fosberg KK, Puentedura E, Schmitz B, Jain TK, Cleland JA. The Effects of Thrust Joint Manipulation on the Resting and Contraction Thickness of Transversus Abdominis in Patients With Low Back Pain: A Randomized Control Trial. J Manipulative Physiol Ther. 2020 May;43(4):339-355. doi: 10.1016/j.jmpt.2019.04.006. Epub 2020 Jul 21. PMID 32709514